CLINICAL TRIAL: NCT01510119
Title: Autophagy Inhibition to Augment Mammilian Target of Rapamycin (mTOR) Inhibition: A Phase I/II Trial of RAD001 and Hydroxychloroquine (HCQ) in Patients With Previously Treated Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: University of Pittsburgh (Other); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 07811
Record Dates: First submitted 2012-01-11; First posted 2012-01-13 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Metastatic Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma | interventions — Hydroxychloroquine; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention - Dose Level 1 (Experimental): RAD001 given 10mg/daily by mouth and 400mg hydroxychloroquine twice daily by mouth. Cycle 1 will include 1 week run-in of RAD001. Following this, both RAD001 and hydroxychloroquine given without interruption. Cycle 1 duration is 35 days; all subsequent cycles are 28 days. RAD001 and hydroxychloroquine continuously administered until progression of disease or unacceptable toxicity.
  Interventions: Drug: Hydroxychloroquine; Drug: RAD001
- Intervention - Dose Level 2 Phase 2 (Experimental): RAD001 given 10mg/daily by mouth and 600mg hydroxychloroquine twice daily by mouth. Cycle 1 will include 1 week run-in of RAD001. Following this, both RAD001 and hydroxychloroquine given without interruption. Cycle 1 duration is 35 days; all subsequent cycles are 28 days. RAD001 and hydroxychloroquine continuously administered until progression of disease or unacceptable toxicity.
  Interventions: Drug: Hydroxychloroquine; Drug: RAD001

INTERVENTIONS:
Drug: Hydroxychloroquine
  Other Names: HCQ
Drug: RAD001
  Other Names: Everolimus; Afinitor

SUMMARY:
This is an open labeled phase I dose escalation study of hydroxychloroquine (HCQ) and RAD001 in patients with advanced renal cell carcinoma followed by a Phase II trial of RAD001 with HCQ. The target population are patients with one to three prior treatments for advanced renal cell carcinoma. In the phase I portion a traditional 3+3 design will be used to determine the maximal tolerated dose and/or recommended phase II dose for HCQ in combination with RAD001 po 10 mg/day.

DETAILED DESCRIPTION:
This protocol describes a multicenter phase I/II trial of RAD001 in combination with hydroxychloroquine (HCQ) (phase I anticipated n=6-12) with a 35 patient phase II trial in patients with previously treated (1-3 prior regimens) advanced renal cell carcinoma. The preclinical rationale for this combination is extensive, the safety of HCQ combination strategies has been established, and effective autophagy pharmacodynamics (PD), and pharmacokinetics (PK) assays are available to guide development. The practical advantage of combination with HCQ is that this drug is off patent, commercially available, and is investigational new drug (IND) exempt. The institutions involved have combined 11 clinical protocols open for accrual involving HCQ, so regulatory approval will be rapid. There are no competing HCQ protocols for advanced renal cell carcinoma. As described in the sample size justification we are setting a high threshold to consider RAD001 + HCQ active since there are many competitors and other potential rational combinations. The 35 patient sample size is designed as a 2 stage phase II trial that will guide the go/no-go decision regarding the conduct of a followup randomized study to definitively prove efficacy. The primary (6 month PFS) and secondary outcomes (response rate, toxicity rates, correlative endpoints) will be analyzed for the entire group, and for patient populations stratified by number of prior therapies. The phase I portion of this trial is anticipated to be short, based on our experience from other HCQ trials. As a safety measure we have included intermediate dose levels which will only be used if there are Dose Limiting Toxicities (DLTs). Since we have seen responses at lower doses of HCQ in other trials, and because frequently over months HCQ dose is lowered from Maximum Tolerated Dose (MTD) doses in many trials because of nausea and anorexia, we would like to have some data on renal cell patients treated at the lower dose levels. If there is activity demonstrated at lower doses, this would be informative for dose modification decisions in patients treated on the dose expansion. The patient population for this trial, including the phase I dose escalation portion is advanced renal cell carcinoma with 1-3 prior treatments.

ELIGIBILITY:
Inclusion Criteria:

* 1 Histological evidence of metastatic renal cell carcinoma that has been previously treated with 1-3 prior regimens
* 2 Phase I only, any number of prior regimens with evidence of progressive disease
* 3 Patients must have at least one measurable site of disease according to RECIST criteria that has not been previously irradiated. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation
* 4 Age 18 years
* 5 Eastern Cooperative Oncology Group (ECOG) performance status £
* 6 Adequate bone marrow function as shown by: absolute neutrophil count (ANC) 1.5 x 109/L, Platelets 100 x 109/L, Hb 9 g/dL
* 7 Adequate liver function as shown by:
* 8 Serum bilirubin 1.5 x upper limit of normal
* 9 ALT and aspartate aminotransferase (AST) 2.5x upper limit of normal ( 5x upper limit of normal in patients with liver metastases)
* 10 international normalized ratio (INR) and PTT 1.5. (Anticoagulation is allowed if target INR 1.5 on a stable dose of warfarin or on a stable dose of anticoagulant for 2 weeks at time of randomization.) Adequate renal function: serum creatinine 2.0 x upper limit of normal or Creatinine Clearance 60 .11 Fasting serum cholesterol 300 mg/dL OR 7.75 mmol/L AND fasting triglycerides 2.5 x upper limit of normal . NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* 12 Signed informed consent

Exclusion Criteria:

.1. Patients currently receiving anticancer therapy or who have received anticancer therapy within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.). To prevent explosive disease progression associated with angiogenic rebound from impacting the results of this study, patients who have received prior antiangiogenic therapy in the form of a small molecule multikinase inhibitor or bevacizumab must be off prior therapy for 1 week and have antiangiogenic therapy-associated adverse events (AEs) resolve to grade 2 before starting study treatment.

* 2 Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery or patients that may require major surgery during the course of the study
* 3 Prior treatment with any investigational drug within the preceding 4 weeks .4 Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* 5 Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* 6 Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* 7 Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin, Stage I resected melanoma, ductal carcinoma in situ, squamous cell carcinoma of the skin, resected, basal cell carcinoma, indolent prostate cancer
* 8 Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* 9 Symptomatic congestive heart failure of New York heart Association Class III or IV
* 10 Unstable angina pectoris, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
* 11 Severely impaired lung function with a previously documented spirometry and diffusing capacity of lung for carbon monoxide that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
* 12 Uncontrolled diabetes as defined by fasting serum glucose 1.5 x ULN
* 13 Active (acute or chronic) or uncontrolled severe infections
* 14 Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* 15 A known history of HIV seropositivity as reported by the patient
* 16 Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* 17 Patients with an active, bleeding diathesis
* 18 Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of RAD001)
* 19 Patients who have received prior treatment with an mammilian target of rapamycin (mTOR) inhibitor (sirolimus, temsirolimus, everolimus).(Phase I prior mTOR inhibitor allowed)
* 20 Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients
* 21 History of noncompliance to medical regimens
* 22 Patients unwilling to or unable to comply with the protocol .23 A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. HBV DNA and HCV RNA polymerase chain reaction testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-04-04 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
PFS | 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Medicine and Dentistry of New Jersey, New Brunswick, New Jersey
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Hillman Cancer Center, Pittsburgh, Pennsylvania